CLINICAL TRIAL: NCT03491085
Title: Study Of The Antibiotic Role In Post Tonsillectomy Complications
Brief Title: Role of Antibiotics Post Tonsillectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ahmedz, principal investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Antibiotics with tonsillectomy
Record Dates: First submitted 2018-03-16; First posted 2018-04-09 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tonsillictomy with antibiotics (Active Comparator)
  Interventions: Drug: Amoxicillin/clavulanate
- tonsillictomy Without Antibiotics (No Intervention)

INTERVENTIONS:
Drug: Amoxicillin/clavulanate — after tonsillectomy half of our patients will receive Amoxicillin /clavulanate for one week and the other half will not receive it.
  Arms: tonsillictomy with antibiotics

SUMMARY:
morbidity after tonsillictomy remains asignificant problem therefore they recommend prophylactic antibiotics to reduce it.in the other hand, the overuse of antimicrobial agents can lead to antimicrobial resistance ,adverse drug events,and unnecessary cost.so,the effectiveness and necessity of antibiotic following tonsillictomy needs to be studied .

ELIGIBILITY:
Inclusion Criteria:

200 patients who are scheduled for tonsillectomy with or without adenoidectomy, and their age are less than 18 years old of either gender will be included in our study

Exclusion Criteria:

* 1-Patients age ≥ 18 years.

  2-Trials in which antibiotics was administrated locally or used in the immediate preoperative period (within seven days before surgery).

  3. Medical comorbidity requiring treatment with antibiotics e.g. Rheumatic heart disease

  4-Patients undergoing the following procedures:
  1. Unilateral tonsillectomy or biopsy.
  2. Tonsillectomy for known carcinoma.
  3. Tonsillectomy in conjunction with palatal surgery.
  4. Hot tonsillectomy for tonsillar abscess

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
compare the morbidity after tonsillectomy between the group which receive antibiotics and the other group which not receive antibiotics | 2 years
  A questionnaire will be given to the parents on discharge to fill in the type of post-tonsillectomy morbidity of main concern including: fever, secondary bleeding, number of days with throat pain and the number of days to resume normal diet, incidence of abdominal pain, nausea & vomiting.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel A, Foden N, Rachmanidou A. Is weekend surgery a risk factor for post-tonsillectomy haemorrhage? J Laryngol Otol. 2016 Aug;130(8):763-7. doi: 10.1017/S0022215116008161. Epub 2016 Jun 13. PMID 27292442